CLINICAL TRIAL: NCT06283979
Title: A Multi-center, Randomized (1:1), Controlled Phase II Trial of STIMULAN VG With Debridement and a Course of Systemic Antibiotics vs Standard of Care (SoC) for the Treatment of Osteomyelitis Associated With Stage IV Pressure Ulcers.
Brief Title: A Randomized Controlled Phase II Trial of STIMULAN VG vs Standard of Care (SoC) for the Treatment of Osteomyelitis Associated With Stage IV Pressure Ulcers.
Acronym: BLADE OPU2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocomposites Ltd (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199723
Expanded Access: NCT06808568 (Available)
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Pressure Ulcer, Stage IV; Osteomyelitis
Keywords: between-group effect size; surgical debridement; ulcer bursectomy; systemic antibiotics
MeSH Terms: conditions — Pressure Ulcer; Osteomyelitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional STIMULAN VG (Experimental): Ulcer bursectomy and debridement and STIMULAN VG insertion into the ulcer cavity.
  Flap/primary closure. Peri-operative antibiotics.
  Interventions: Combination Product: STIMULAN VG; Procedure: Standard of Care
- Standard of Care (SoC) (Active Comparator): Ulcer bursectomy, debridement and flap/primary closure. Peri-operative antibiotics.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Combination Product: STIMULAN VG — Insertion of STIMULAN VG into the ulcer cavity prior to flap/primary closure.
  Arms: Interventional STIMULAN VG
Procedure: Standard of Care — Standard of Care. Ulcer bursectomy, debridement and flap/primary closure. Peri-operative antibiotics.

SUMMARY:
The purpose of this trial is to assess the safety, tolerability and between-group effect size of STIMULAN VG (with debridement) and a course of systemic antibiotics to standard of care (debridement and systemic antibiotics only) for the treatment of osteomyelitis associated stage IV pressure ulcers.

DETAILED DESCRIPTION:
The trial is an open-label, multi-center, randomized (1:1), controlled phase 2 trial in patients diagnosed with stage IV pressure ulcers.

ELIGIBILITY:
In order to be eligible to participate in this study, subjects must meet all of the following criteria:

1. Presenting with a Stage IV pressure ulcer requiring treatment of excision, bony debridement and flap coverage/primary closure.
2. Operative candidate for flap surgery or primary closure.
3. Presence of focal osteomyelitis as suggested by imaging to show extent of infection. Acceptable imaging techniques are Magnetic Resonance Imaging or CT scan.
4. Adults ≥ 18 years in age at the time of treatment.
5. Psychosocially, mentally, and physically able to fully comply with this protocol, including adhering to scheduled visits, treatment plan, completing forms, and other study procedures.
6. Ability of the subject or legal authorized representative to provide voluntary, signed and dated informed consent prior to any study-related procedures.

Subjects who meet any of the following criteria will be excluded from participating in this study:

1. Reasons contributing to pressure ulcer cannot be addressed.
2. Severe immunological compromised patients as determined by the clinician.
3. Patients with diffuse or widespread pelvic osteomyelitis that is not amenable to adequate margins for debridement.
4. Patients presenting with head pressure ulcers.
5. Current or recent history (within last 2 years) of active substance abuse (e.g., recreational drugs, narcotics, or alcohol) that in the judgement of the investigator, may compromise the participant's safety/recovery or ability to follow the trial procedures.
6. Current smoker.
7. Diabetic patient with Hba1C level above 9.
8. Allergy to any component of the investigational product, such as calcium sulfate, glycopeptide antibiotics (Vancomycin), or aminoglycoside antibiotics (Gentamicin).
9. Concurrent involvement in a study of another investigational product.
10. Pregnant or planning to become pregnant during study period.
11. Flexion contractures where patient cannot passively get full extension.
12. Uncontrolled muscle spasms.
13. Unable to comply with bedrest restriction or offloading requirements
14. Unable to provide consent.
15. Fecal or urinary incontinence with contamination of the wound.
16. Lower extremity pressure ulcer location that is vascularly compromised as defined by an Ankle Brachial Index ≤ 0.7 mm Hg OR toe brachial index ≤ 0.6 mm OR toe pressure ≤ 40 mm Hg OR transcutaneous oximetry ≤ 40 mm Hg *
17. Investigator considers the participant to be clinically malnourished.
18. Any conditions with known hypercalcemia (> 10.3 mg/dl) or posing a significant risk for developing hypercalcemia (i.e., Hyperparathyroidism).
19. Investigator believes trial participation may compromise safety of the participant or trial results.

    * Patients presenting with lower extremity pressure ulcers that are vascularly compromised can be rescreened followed successful revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Individual patient success and findings at the 8 week follow-up visit | 8 week
  An individual patient treatment will be considered a success if there is complete wound closure and healing at the surgical site at two consecutive visits 2 weeks apart.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Advanced Foot Care, LLC, Phoenix, Arizona
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Hospital - Long Island Clinical Research Center, Mineola, New York
  - University of Pittsburgh, McGowan Institute for Regenerative Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No